CLINICAL TRIAL: NCT04928495
Title: Clinical, Control, Double-blind, Randomized Experimentation With N-acetylcysteine and Bromhexine for COVID-19
Brief Title: Clinical Trial With N-acetylcysteine and Bromhexine for COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Ceara (Other)
Collaborators: Paulista School of Medicine-EPM, UNIFESP (Unknown); Health Surveillance Secretariat - SVS (Unknown); Central Laboratory of Public Health of Ceara - LACEN-CE (Unknown); Leonardo da Vinci Hospital - HLV (Unknown); São José Hospital for Infectious Diseases - HSJ (Unknown); Ceará Health Secretariat - SESA (Unknown); Municipal Health Secretary - SMS-Fortaleza (Unknown)
Responsible Party: Principal Investigator, Aldo Ângelo Moreira Lima, Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVANTI-C19
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: N-acetylcysteine; Bromhexine; COVID-19; Clinical trial
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid; Acetylcysteine; Bromhexine

STUDY DESIGN:
Intervention Model Description: (1) Placebo control; (2) N-acetylcysteine treatment (NAC); and (3) NAC + Bromhexine treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical trial will be masked by participant, care provider, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Placebo Comparator): Control placebo (Vitamin C - 500mg / day, for 10 days)
  Interventions: Drug: Vitamin C
- Treatment group 2 (Active Comparator): N-acetylcysteine (NAC; 1800 mg / day, for 10 days)
  Interventions: Drug: N-acetylcysteine (NAC)
- Treatment group 3 (Active Comparator): NAC (1800 mg / day) + bromhexine-BMX (32 mg / day for 10 days)
  Interventions: Drug: NAC + Bromhexine (BMX)

INTERVENTIONS:
Drug: Vitamin C — Vitamin C 500 mg / day for ten days
  Arms: Treatment group 1
Drug: N-acetylcysteine (NAC) — N-acetylcysteine 1800 mg / day for ten days.
  Arms: Treatment group 2
Drug: NAC + Bromhexine (BMX) — NAC + Bromhexine (BMX) 32 mg / day for ten days.
  Arms: Treatment group 3

SUMMARY:
Clinical, control, double-blind, randomized experimentation with N-acetylcysteine and bromhexine for COVID-19.

DETAILED DESCRIPTION:
Several therapeutic agents have been evaluated for the treatment of COVID-19, but only one, the antiviral drug called remdesivir administered intravenously, has shown to be effective in shortening the duration of the disease by 26.7% in critically ill patients. This proposal has the primary objective (1) to determine the effect of N-acetylcysteine (NAC; reducing substance and complementary viral intercepting action) and combination of NAC + bromhexine (BMX; viral protease inhibitor), on the clinical duration of COVID-19 evaluated on the 7th. day of outpatient follow-up, observing the score of clinical signs and symptoms of the disease. The study has as secondary objectives: (2) to assess the change in viral load by RT-qPCR of SARS-CoV-2 between the 1st, 7th, and 14th. days of the experimental protocol; (3) determine the action of NAC and BMX + NAC on the immune response using the rapid ELISA test (IgM / IgG) to be performed on the 14th. monitoring day of the experimental protocol; and (4) Assess the effect of NAC and BMX + NAC on the change in the serum level of inflammation biomarkers and reducing substances (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF- α, MCP-1, IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I, PCR and procalcitonin; glutathione peroxidase-GPx; superoxide dismutase-SOD and catalase-CAT) of patients collected on the 1st. and 14 o. study days. The study will be a prospective, double-blind, placebo control and randomized clinical trial of a total of 219 patients, 73 for each treatment group, with mild to moderate disease, equal to or above 18 years of age, with clinical signs and symptoms. of COVID-19 and certified by the RT-qPCR test for the detection of SARS-CoV-2 viral load. The study will be carried out using the Surveillance, Service and Research Network - REVAP-C19, NUBIMED, FAMED, UFC, Fortaleza, CE in order to facilitate the efficiency of patients' entry into the study. The random groups of treatments will be: (1) Placebo control (Vitamin C - 500 mg / day, for 10 days); (2) N-acetylcysteine (NAC; 1800 mg / day, for 10 days); and (3) NAC (1800 mg / day, for 10 days) + Bromhexine Hydrochloride (BMX; 32 mg / day, for 10 days). The study has the perspective of evaluating the effectiveness of NAC alone or combined with BMX in the duration of the clinical score of mild to moderate cases of COVID-19. The study will also assess secondary parameters such as the effect of drugs on changing viral load, immune response, and changing the inflammatory reaction and reducing substances in the plasma of the study patients. In this sense, the trial plans to minimize the evolution of the disease to severe cases, thus alleviating the collapse of the health system and minimizing the social, economic and health disorders of the pandemic by SARS-CoV-2.

ELIGIBILITY:
The inclusion criteria will be:

1. patients with clinical signs and symptoms of COVID-19; and
2. patients over 18 years and below 60 years of age.

The exclusion criteria will be:

1. participate in another clinical intervention study;
2. you have a disease or other medical condition that prevents you from using the medications for this intervention;
3. patient incapable of ingesting, retaining and absorbing the intervention medications; and (d) is mentally disabled.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 219 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-06-09 (Estimated)

PRIMARY OUTCOMES:
The time to recovery, defined at day 7 days follow up after enrollment, on which a patient met the criteria for category 1 or 2 on the four-category ordinal scale. [Time Frame: Day 7 follow up after enrollment.] | Day 7
  The categories are as follows: 1 - No signals and symptoms; 2 - One signal or symptom; 3 - Two signals or symptoms; 4 - Three or more signals or symptoms.

SECONDARY OUTCOMES:
SARS-CoV-2 RNA viral load measurements change. [ Time Frame: Change between Day 1 and Day 7 follow up after enrollment. ] | Day 1 and Day 7
  Molecular diagnostic analyzes will be done by Real-Time PCR (qPCR) based on official guidelines determined by the American CDC (CDC-006-00019, Revision: 03; https://www.fda.gov/media/134922/download). The nasopharyngeal swab samples collected (Covid-19 test) will proceed to the nucleic acid isolation (NuAc). All qPCR reactions will be by uniplex diagnosis. Results will be reported in copies of RNA / ml.
Proportion of patients with qualitative serum IgM / IgG. [ Time Frame: Proportion of positive patients at Day 7 for IgM / IgG (N; %). ] | Day 7
  The IgM / IgG immune response to SARS-CoV-2 will be qualitative measure using rapid diagnostic test provide by Eco Diagnóstica (Nova Lima, MG, Brazil).
Biomarkers (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF-α, MCP-1, IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I, CRP and procalcitonin) measurements change. [ Time Frame: Change between Day 1 and Day 14 follow up after enrollment. ] | Day 1 and Day 14.
  We will use the Luminex XMAP Technology (MAGPIX® System, Merck Co., Kenilworth, NJ) which includes the simultaneous analysis, in the same plasma sample (volume of 25 uL), of a panel of protein markers of pro and anti-inflammatory activity (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF-α, MCP-1, IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I). Specific antibodies covalently linked to the carboxylated microspheres containing different specific fluorochromes will be used. Standard curves will be constructed for each protein and then their quantification. Results will be reported in pg / mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Núcleo de Biomedicina - NUBIMED, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided